CLINICAL TRIAL: NCT06025409
Title: A Phase III Clinical Trial to Evaluate the Efficacy and Safety of DWJ108J in Patients With Central Precocious Puberty : A Single-arm, Open-label, Multi-center, Prospective Study
Brief Title: Evaluate the Efficacy and Safety of DWJ108J
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ108J301
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Leuprorelin (Experimental): Participants with body weight greater than or equal to (≥) 20 kilogram (kg) will receive the recommended dose of leuprorelin 11.25 milligram (mg), injection, subcutaneously, once every 3 months for 6 months. Participants with body weight less than (<) 20 kg will receive leuprorelin 5.625 mg, injection, subcutaneously, once every 3 months for 6 months.
  Interventions: Drug: Leuprolide Acetate 11.25 MG/ML

INTERVENTIONS:
Drug: Leuprolide Acetate 11.25 MG/ML — Subcutaneous injection

SUMMARY:
This study aims to evaluate the efficacy and safety of DWJ108J (Leuprorelin acetate 11.25 mg) in patients with central precocious puberty.

DETAILED DESCRIPTION:
The drug in this study is called leuprorelin. It is administered as a 3 month subcutaneous depot injection. Leuprorelin is used to treat children who have Central Precocious Puberty. This study will look at whether leuprorelin can stop early Central Precocious Puberty.

ELIGIBILITY:
Inclusion Criteria:

1. Exhibited pubertal response of LH (peak ≥ 5 IU/L) during GnRH stimulation test at screening
2. Diagnosis of central precocious puberty
3. For boys, those under 10 years old and for girls, those under 9 years old, based on Visit 2 (Enrollment), with Tanner Stage 2 or above
4. Difference between bone age (Greulich and Pyle method) and chronological age ≥ 1 year
5. In cases where the legal guardian of the child listened to the explanation of this clinical trial and provided written consent

Exclusion Criteria:

1. Following conditions at Visit 1(Screening) :

   Conditions related to pseudo precocious puberty, Incomplete precocious puberty, Dysfunction of pituitary, adrenal, thyroid, or reproductive glands, Growth disorders or bone diseases that could affect bone growth, Brain tumor, Pituitary adenoma
2. requires treatment within 6 months of receiving a registration number during the trial period that could affect the hypothalamic-pituitary-gonadal axis
3. Prior treatment with GnRH analogues
4. Hypersensitive to the investigational drug for this clinical trial or GnRH analogues
5. Prior or current therapy with growth hormone
6. has taken the following medications within 8 weeks of Visit 1 (Screening): Sex hormone medications, Sex hormone antagonists, Steroids (local application is allowed; oral formulations are not allowed if taken within 3 days continuously, and use within 2 weeks of screening is prohibited), Herbal medicine
7. Meets the following criteria based on screening test results:

   AST, ALT levels exceed twice the upper limit of normal, Creatinine levels exceed 1.5 times the upper limit of normal, Bone age is above 11.5 years
8. Any other medical condition or serious intercurrent illness that, in the opinion of the Investigator, may make it undesirable for the subject to participate in the study

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Suppression of Peak-Stimulated Luteinizing Hormone at 6 Months. | 6 months
  Luteinizing Hormone (LH) suppression is defined as peak-stimulated LH ≤ 3 IU/L.

SECONDARY OUTCOMES:
Percentage of Participants With Suppression of Peak-Stimulated Luteinizing Hormone at 3 Months. | 3 months
  Luteinizing Hormone (LH) suppression is defined as peak-stimulated LH ≤ 3 IU/L.
Average LH and FSH concentrations at each time point, and the changes from baseline levels before administration. | Baseline, 3 and 6 months
  Average LH and FSH concentrations at each time point, and the changes from baseline levels before administration.
Average LH peak and FSH peak through GnRH stimulation test at 3 and 6 months after administration, and the changes in each time point compared to before administration | 3 and 6 months
  Average LH peak and FSH peak through GnRH stimulation test at 3 and 6 months after administration, and the changes in each time point compared to before administration
Average concentrations of Estradiol or Testosterone at each time point, and the respective changes compared to before administration. | Baseline, 3 and 6 months
  Average concentrations of Estradiol or Testosterone at each time point, and the respective changes compared to before administration.
Average bone age/chronological age ratio at 6 months after administration, and the changes compared to before administration. | 6 months
  Average bone age/chronological age ratio at 6 months after administration, and the changes compared to before administration.
Average Tanner Stage at 6 months after administration, and the changes compared to before administration. | 6 months
  Average Tanner Stage at 6 months after administration, and the changes compared to before administration.
Average growth velocity (cm/year, annualized height velocity) at 6 months after administration, and the changes compared to before administration. | 6 months
  Average growth velocity (cm/year, annualized height velocity) at 6 months after administration, and the changes compared to before administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Soong Hwang, MD. PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University medical center, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No